CLINICAL TRIAL: NCT04172168
Title: Clinical Characteristics of Left Ventricular Free-wall Ruptrue After Acute Myocardial Infarction
Brief Title: Left Ventricular Free-wall Ruptrue After Acute Myocardial Infarction (LVFR-AMI)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xiamen Cardiovascular Hospital, Xiamen University (Other)
Responsible Party: Principal Investigator, Yan Wang, President, Xiamen Cardiovascular Hospital, Xiamen University
Other Study IDs: 9215443689
Record Dates: First submitted 2019-11-18; First posted 2019-11-21 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Acute Myocardial Infarction
Keywords: Left Ventricular Free-wall Ruptrue; Acute myocardial infarction; Coronary angiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Heart rupture: Include left ventricular free-wall ruptrue after AMI
  Interventions: Diagnostic Test: Heart rupture
- Non heart rupture: AMI with non heart rupture

INTERVENTIONS:
Diagnostic Test: Heart rupture — Left ventricular free-wall ruptrue after AMI
  Groups: Heart rupture

SUMMARY:
The Left Ventricular Free-wall Ruptrue (LVFR) is a serious complication caused high mortality.

DETAILED DESCRIPTION:
The actual mortality of LVFR is close to 100%. Despite the mortality rate for LVFR has been decreasing with the development of reperfusion therapy, the serious complication remains a difficult challenge. The coronary anatomy distribution associated with LVFR has an interesting phenomenon. From the perspective of different coronary distribution, we can better known the risk factors related to LVFR.

ELIGIBILITY:
Inclusion Criteria:

* Patients be admitted for acute myocardial infarction (STEMI or NSTEMI)

Exclusion Criteria:

* Non-cardiovascular comorbidity for AMI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population of acute myocardial infarction (STEMI or NSTEMI) patients.
Sampling Method: Non-Probability Sample
Enrollment: 17568 (Estimated)
Dates: Start 2011-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Rate of heart ruputre | Mortality 30 days
  Left Ventricular Free-wall Ruptrue

SECONDARY OUTCOMES:
Rate of cardiogenic shock | Hospitalization 30 days
  Cardiogenic shock After AMI
Rate of cardiac arrest | Hospitalization 30 days
  Cardiac arrest After AMI

CONTACTS AND LOCATIONS:
Overall Officials: Yan Wang, PhD, Study Chair — Cardiovascular Hospital, Xiamen University
Locations (1):
- Xiamen Cardiovascular Hospital Xiamen University, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No